CLINICAL TRIAL: NCT03691961
Title: Therapeutic Drug Monitoring of Corticosteroids/β2-agonists in Hair in Asthmatic Patients: an Open-label Feasibility Study
Brief Title: Corticosteroids/β2-agonists in Hair in Asthmatic Patients (CorticHair)
Acronym: CorticHair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017047F
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Half of the patients is enrolled in each group according to the individual dose decided by the clinician in charge as the optimal dose to treat the disease. The optimized dose to treat the disease is decided independently of the participation to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium dose of Symbicort Turbuhaler® (Experimental): The population is asthmatic patients meeting the inclusion and exclusion criteria for whom the optimized total daily dose to treat the disease is ≥400 to 800 µg budesonide of budesonide/formoterol Symbicort Turbuhaler®.
  Hair sampling after 4 months treatment.
  Analysis of hair's drug concentrations.
  Interventions: Other: Hair sampling; Diagnostic Test: Hair's drug concentrations
- High dose of Symbicort Turbuhaler® (Experimental): The population is asthmatic patients meeting the inclusion and exclusion criteria for whom the optimized total daily dose to treat the disease is ≥800 µg budesonide of budesonide/formoterol Symbicort TurbuhalerTurbuhaler®.
  Hair sampling after 4 months treatment.
  Analysis of hair's drug concentrations.
  Interventions: Other: Hair sampling; Diagnostic Test: Hair's drug concentrations

INTERVENTIONS:
Other: Hair sampling — After 4 months of treatment, a strand of hair from the vertex posterior region of the scalp about the width of a thin pencil and with a length equal to or greater than 3 cm will be cut.
Diagnostic Test: Hair's drug concentrations — The hair's concentrations of budesonide/formoterol is analysed with mass spectrometry.

SUMMARY:
This feasibility study will be open-label with two dose groups: patients receiving budesonide/formoterol Turbuhaler® at a total daily dose [400 to 800 µg[ (group 1) and patients receiving a total daily dose ≥800 µg/day (group 2) to investigate whether there is a relationship between dose and hair concentration.

The objective of this feasibility study is to determine if the product administered to the patient is detectable and quantifiable in hair in order to have a mean to monitor adherence to the treatment. This study does not in any way evaluate the efficacy or safety of the medicinal product, which will be used in accordance with its marketing authorization.

DETAILED DESCRIPTION:
Asthma affects 3-10% of the European population and is a heterogeneous disease in its clinical manifestations and also in its response to treatment. Since therapy is often started at young age and given over many years, with adjustments made on disease control, long-term adherence and efficacy are particular concerns.

Adherence to inhaled controller medications is a major challenge to obtain disease control and to avoid serious asthma flare-ups or unnecessary treatment stepping up. In addition to adherence concerns, poor asthma control may also be the consequence of a poor inhalation technique and the resulting insufficient drug exposure.

To overcome adherence issues, patients are encouraged to self-manage their disease and the use of new technologies such as inhaler reminders, electronic devices and/or smartphone applications may be helpful. Although there is a margin to improve and monitor adherence, assessing the efficiency of the inhalation technique in daily routine and its consequences in terms of drug exposure is much harder.

The traditional monitoring of pharmacological therapies involves therapeutic drug monitoring, i.e. the measure of drug concentration in plasma. But drugs concentration in plasma most only reflect the quantity of drug in the body in the last 24-48 hrs only. Hence, therapeutic drug monitoring is not used for inhaled asthma treatments, in part because of the limited interest in assessing only a 24-48 hrs exposure and of the very low plasma concentrations which are very challenging to measure.

Since drugs present in the bloodstream also reach and stay in the forming hair where their concentrations can be measured and interpreted as an overall chronic exposure, hair analysis could become a valuable tool in the monitoring of inhaled asthma treatments, with the use of very specific mass spectrometry techniques and of the most sensitive last-generation mass spectrometers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedure
* Outpatients with asthma, of either gender, aged ≥18 and <50 years at visit 1
* Controlled or partly controlled asthma according to the Global Initiative for Asthma (GINA) guideline
* Receiving a constant daily dose ≥400 µg budesonide of budesonide/formoterol Turbuhaler® for more than 2 months
* No treatment step-down is planned in the 3 next months
* ACQ (Asthma Control Questionnaire) score ≤ 1.50
* Patient with healthcare insurance

Exclusion Criteria:

* Pregnant women or women wishing to become pregnant in the next 3 months
* Patients with body mass index (BMI) <18 or >30
* Patients with known kidney or liver disease (creatinine clearance < 60 mL/min/1.73 m² or alanine aminotransferase (ALAT) > 5N)
* Smokers or former smokers < 3 years
* Patients with simultaneous asthma and chronic obstructive pulmonary disease (COPD) (or defined as having asthma-COPD overlap syndrome)
* Other budesonide- or formoterol-containing drugs (e.g Foradil®, Rhinocort®, Mikicort®, Entocort®…)
* CYP3A4 inducers (systemic corticosteroid, rifampicin, phenobarbital, carbamazepine…)
* CYP3A4 inhibitors (macrolides, azole antifungals, valproic acid, amiodarone, fluoxetine)
* Hair treatment (coloration, bleaching, perming…)
* Hairless patients, hair implants or hair extensions
* Length of hair from the vertex posterior region < 5 cm or planning to cut hair from this region shorter than 5 cm in the next 4 months
* Patient deprived of liberty by judicial or administrative decision
* Major protected by law

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Budesonide/formoterol hair concentrations (active substance and metabolites) | 4 months
  After 4 months of treatment, the hair's concentrations of budesonide/formoterol is analyzed with mass spectrometry.

SECONDARY OUTCOMES:
Budesonide/formoterol concentration in three 1-cm hair segments (active substance and metabolites) | 4 months
  After 4 months of treatment, the concentrations of budesonide/formoterol in three 1-cm hair segments is analyzed with mass spectrometry.
Budesonide/formoterol hair's concentration compared to the daily observance. | 4 months
  Patient cumulative dose is estimated from daily observance recorded by the patient in the observance record.
Correlation between budesonide/formoterol hair concentrations, forced expiratory volume in 1 second (FEV1), and asthma control questionnaire (ACQ) | 4 months
  FEV1 (measured according to a standardized spirometry technique), and ACQ (patients with a score below 1.0 will have adequately controlled asthma and above 1.0 their asthma will not be well controlled) are collected at the inclusion visit and the 4 months visit

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Grassin-Delyle, Dr, Study Director — University Versailles Saint Quentin / Foch Hospital
Locations (1):
- Foch Hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Jahdali H, Ahmed A, Al-Harbi A, Khan M, Baharoon S, Bin Salih S, Halwani R, Al-Muhsen S. Improper inhaler technique is associated with poor asthma control and frequent emergency department visits. Allergy Asthma Clin Immunol. 2013 Mar 6;9(1):8. doi: 10.1186/1710-1492-9-8. PMID 23510684
- [Background] Alonso L, Fuchs E. The hair cycle. J Cell Sci. 2006 Feb 1;119(Pt 3):391-3. doi: 10.1242/jcs.02793. No abstract available. PMID 16443746
- [Background] Alvarez JC, Abe E, Etting I, Le Guen M, Devillier P, Grassin-Delyle S. Quantification of remifentanil and propofol in human plasma: a LC-MS/MS assay validated according to the EMA guideline. Bioanalysis. 2015;7(13):1675-84. doi: 10.4155/bio.15.89. PMID 26226314
- [Background] Alvarez JC, Charbit B, Grassin-Delyle S, Demolis JL, Funck-Brentano C, Abe E. Human plasma quantification of droperidol and ondansetron used in preventing postoperative nausea and vomiting with a LC/ESI/MS/MS method. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Jan 15;879(2):186-90. doi: 10.1016/j.jchromb.2010.12.001. Epub 2010 Dec 16. PMID 21185793
- [Background] Auchus RJ. Steroid assays and endocrinology: best practices for basic scientists. Endocrinology. 2014 Jun;155(6):2049-51. doi: 10.1210/en.2014-7534. No abstract available. PMID 24837046
- [Background] Baxi SM, Greenblatt RM, Bacchetti P, Jin C, French AL, Keller MJ, Augenbraun MH, Gange SJ, Liu C, Mack WJ, Gandhi M; Women's Interagency HIV Study (WIHS). Nevirapine Concentration in Hair Samples Is a Strong Predictor of Virologic Suppression in a Prospective Cohort of HIV-Infected Patients. PLoS One. 2015 Jun 8;10(6):e0129100. doi: 10.1371/journal.pone.0129100. eCollection 2015. PMID 26053176
- [Background] Bevalot F, Gaillard Y, Lhermitte MA, Pepin G. Analysis of corticosteroids in hair by liquid chromatography-electrospray ionization mass spectrometry. J Chromatogr B Biomed Sci Appl. 2000 Apr 14;740(2):227-36. doi: 10.1016/s0378-4347(00)00085-2. PMID 10821409
- [Background] Borges NC, Astigarraga RB, Sverdloff CE, Borges BC, Paiva TR, Galvinas PR, Moreno RA. Budesonide quantification by HPLC coupled to atmospheric pressure photoionization (APPI) tandem mass spectrometry. Application to a comparative systemic bioavailability of two budesonide formulations in healthy volunteers. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Feb 1;879(3-4):236-42. doi: 10.1016/j.jchromb.2010.12.003. Epub 2010 Dec 13. PMID 21233029
- [Background] Buscher BA, Jagfeldt H, Sandman H, Brust-van Schaik R, van Schaik F, Brull LP. The determination of budesonide and fluticasone in human sputum samples collected from COPD patients using LC-MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2012 Jan 1;880(1):6-11. doi: 10.1016/j.jchromb.2011.10.029. Epub 2011 Nov 16. PMID 22169057
- [Background] Capron A, Antunes MV, Wagner SC, Mattevi VS, Vieira N, Leite R, Reginato F, Capra M, Fogliatto L, Wallemacq P, Linden R. First report of imatinib measurement in hair: Method development and preliminary evaluation of the relation between hair and plasma concentrations with therapeutic response in chronic myeloid leukemia. Clin Chim Acta. 2016 Jan 30;453:42-7. doi: 10.1016/j.cca.2015.11.032. Epub 2015 Dec 3. PMID 26657979
- [Background] Chalmers GW, Macleod KJ, Little SA, Thomson LJ, McSharry CP, Thomson NC. Influence of cigarette smoking on inhaled corticosteroid treatment in mild asthma. Thorax. 2002 Mar;57(3):226-30. doi: 10.1136/thorax.57.3.226. PMID 11867826
- [Background] Chèze, M. and Gaulier, J.-M. (2014). Chapter 8 - Drugs Involved in Drug-Facilitated Crimes (DFC): Analytical Aspects: 2-Hair A2 - Kintz, Pascal. Toxicological Aspects of Drug-Facilitated Crimes. Oxford, Academic Press: 181-222.
- [Background] Choi HI, Choi GI, Kim EK, Choi YJ, Sohn KC, Lee Y, Kim CD, Yoon TJ, Sohn HJ, Han SH, Kim S, Lee JH, Lee YH. Hair greying is associated with active hair growth. Br J Dermatol. 2011 Dec;165(6):1183-9. doi: 10.1111/j.1365-2133.2011.10625.x. PMID 21916889
- [Background] Cirimele V, Kintz P, Dumestre V, Goulle JP, Ludes B. Identification of ten corticosteroids in human hair by liquid chromatography-ionspray mass spectrometry. Forensic Sci Int. 2000 Jan 10;107(1-3):381-8. doi: 10.1016/s0379-0738(99)00180-2. PMID 10689588
- [Background] Cirimele V, Tracqui A, Kintz P, Ludes B. First identification of prednisone in human hair by liquid chromatography-ionspray mass spectrometry. J Anal Toxicol. 1999 May-Jun;23(3):225-6. doi: 10.1093/jat/23.3.225. No abstract available. PMID 10369335
- [Background] Cochrane MG, Bala MV, Downs KE, Mauskopf J, Ben-Joseph RH. Inhaled corticosteroids for asthma therapy: patient compliance, devices, and inhalation technique. Chest. 2000 Feb;117(2):542-50. doi: 10.1378/chest.117.2.542. PMID 10669701
- [Background] Cone EJ. Mechanisms of drug incorporation into hair. Ther Drug Monit. 1996 Aug;18(4):438-43. doi: 10.1097/00007691-199608000-00022. PMID 8857565
- [Background] Cooper GA, Kronstrand R, Kintz P; Society of Hair Testing. Society of Hair Testing guidelines for drug testing in hair. Forensic Sci Int. 2012 May 10;218(1-3):20-4. doi: 10.1016/j.forsciint.2011.10.024. Epub 2011 Nov 15. PMID 22088946
- [Background] Cuypers E, Flinders B, Bosman IJ, Lusthof KJ, Van Asten AC, Tytgat J, Heeren RMA. Hydrogen peroxide reactions on cocaine in hair using imaging mass spectrometry. Forensic Sci Int. 2014 Sep;242:103-110. doi: 10.1016/j.forsciint.2014.06.035. Epub 2014 Jul 7. PMID 25047217
- [Background] Dalby C, Polanowski T, Larsson T, Borgstrom L, Edsbacker S, Harrison TW. The bioavailability and airway clearance of the steroid component of budesonide/formoterol and salmeterol/fluticasone after inhaled administration in patients with COPD and healthy subjects: a randomized controlled trial. Respir Res. 2009 Oct 31;10(1):104. doi: 10.1186/1465-9921-10-104. PMID 19878590
- [Background] DAVIS BK. Phases of the hair-growth cycle. Nature. 1962 May 19;194:694. doi: 10.1038/194694a0. No abstract available. PMID 13883875
- [Background] Deventer K, Mikulcikova P, Van Hoecke H, Van Eenoo P, Delbeke FT. Detection of budesonide in human urine after inhalation by liquid chromatography-mass spectrometry. J Pharm Biomed Anal. 2006 Oct 11;42(4):474-9. doi: 10.1016/j.jpba.2006.05.016. Epub 2006 Jul 12. PMID 16842962
- [Background] Deventer K, Pozo OJ, Delbeke FT, Van Eenoo P. Quantitative detection of inhaled formoterol in human urine and relevance to doping control analysis. Drug Test Anal. 2012 Jun;4(6):449-54. doi: 10.1002/dta.418. Epub 2012 Mar 22. PMID 22447497
- [Background] Dimova H, Wang Y, Pommery S, Moellmann H, Hochhaus G. SPE/RIA vs LC/MS for measurement of low levels of budesonide in plasma. Biomed Chromatogr. 2003 Jan;17(1):14-20. doi: 10.1002/bmc.204. PMID 12583000
- [Background] Duvivier WF, Peeters RJ, van Beek TA, Nielen MW. Evidence based decontamination protocols for the removal of external Delta9-tetrahydrocannabinol (THC) from contaminated hair. Forensic Sci Int. 2016 Feb;259:110-8. doi: 10.1016/j.forsciint.2015.12.014. Epub 2015 Dec 19. PMID 26773221
- [Background] Fabresse, N. (2015). Mise au point et validation d'une méthode de dosage des anabolisants stéroïdiens dans le sang et les cheveux par spectrométrie de masse haute résolution Orbitrap Application à deux cas médico-légaux, http://www.sudoc.fr/188207155: 93.
- [Background] Fabresse N, Grassin-Delyle S, Etting I, Alvarez JC. Detection and quantification of 12 anabolic steroids and analogs in human whole blood and 20 in hair using LC-HRMS/MS: application to real cases. Int J Legal Med. 2017 Jul;131(4):989-999. doi: 10.1007/s00414-017-1552-3. Epub 2017 Feb 24. PMID 28236045
- [Background] FDA.
- [Background] Foster JM, Usherwood T, Smith L, Sawyer SM, Xuan W, Rand CS, Reddel HK. Inhaler reminders improve adherence with controller treatment in primary care patients with asthma. J Allergy Clin Immunol. 2014 Dec;134(6):1260-1268.e3. doi: 10.1016/j.jaci.2014.05.041. Epub 2014 Jul 22. PMID 25062783
- [Background] Gaillard Y, Vayssette F, Pepin G. Compared interest between hair analysis and urinalysis in doping controls. Results for amphetamines, corticosteroids and anabolic steroids in racing cyclists. Forensic Sci Int. 2000 Jan 10;107(1-3):361-79. doi: 10.1016/s0379-0738(99)00179-6. PMID 10689587
- [Background] Gamble J, Stevenson M, McClean E, Heaney LG. The prevalence of nonadherence in difficult asthma. Am J Respir Crit Care Med. 2009 Nov 1;180(9):817-22. doi: 10.1164/rccm.200902-0166OC. Epub 2009 Jul 30. PMID 19644048
- [Background] Gandhi M, Ameli N, Bacchetti P, Anastos K, Gange SJ, Minkoff H, Young M, Milam J, Cohen MH, Sharp GB, Huang Y, Greenblatt RM. Atazanavir concentration in hair is the strongest predictor of outcomes on antiretroviral therapy. Clin Infect Dis. 2011 May;52(10):1267-75. doi: 10.1093/cid/cir131. PMID 21507924
- [Background] Gandhi M, Greenblatt RM, Bacchetti P, Jin C, Huang Y, Anastos K, Cohen M, Dehovitz JA, Sharp GB, Gange SJ, Liu C, Hanson SC, Aouizerat B; Women's Interagency HIV Study. A single-nucleotide polymorphism in CYP2B6 leads to >3-fold increases in efavirenz concentrations in plasma and hair among HIV-infected women. J Infect Dis. 2012 Nov;206(9):1453-61. doi: 10.1093/infdis/jis508. Epub 2012 Aug 20. PMID 22927450
- [Background] Shen HH, Du XF, Ying SM. [Comparison of Chinese guideline for asthma managment and prevention (2016 update) and global initiative for asthma (2017 update)]. Zhonghua Jie He He Hu Xi Za Zhi. 2018 Mar 12;41(3):166-168. doi: 10.3760/cma.j.issn.1001-0939.2018.03.003. No abstract available. Chinese. PMID 29518845
- [Background] Grassin Delyle S, Abe E, Batisse A, Tremey B, Fischler M, Devillier P, Alvarez JC. A validated assay for the quantitative analysis of tranexamic acid in human serum by liquid chromatography coupled with electrospray ionization mass spectrometry. Clin Chim Acta. 2010 Mar;411(5-6):438-43. doi: 10.1016/j.cca.2010.01.005. Epub 2010 Jan 11. PMID 20064499
- [Background] Grassin Delyle S, Abe E, Devillier P, Alvarez JC. Determination of rimonabant in human plasma and hair by liquid chromatography-mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2008 Sep 1;872(1-2):115-20. doi: 10.1016/j.jchromb.2008.07.041. Epub 2008 Aug 5. PMID 18707925
- [Background] Handelsman DJ, Wartofsky L. Requirement for mass spectrometry sex steroid assays in the Journal of Clinical Endocrinology and Metabolism. J Clin Endocrinol Metab. 2013 Oct;98(10):3971-3. doi: 10.1210/jc.2013-3375. No abstract available. PMID 24098015
- [Background] He G, Lu J, Wang X, Xu Y, Wu Y, Dong Y, Shen L, He Z, Zhao J, Yuan H. An improved liquid chromatography-tandem mass spectrometric method to quantify formoterol in human urine. J Chromatogr Sci. 2014 Sep;52(8):848-51. doi: 10.1093/chromsci/bmt127. Epub 2013 Sep 12. PMID 24029618
- [Background] Hoelzle C, Scheufler F, Uhl M, Sachs H, Thieme D. Application of discriminant analysis to differentiate between incorporation of cocaine and its congeners into hair and contamination. Forensic Sci Int. 2008 Mar 21;176(1):13-8. doi: 10.1016/j.forsciint.2007.07.020. Epub 2007 Dec 11. PMID 18063333
- [Background] Josefsson M, Sabanovic A. Sample preparation on polymeric solid phase extraction sorbents for liquid chromatographic-tandem mass spectrometric analysis of human whole blood--a study on a number of beta-agonists and beta-antagonists. J Chromatogr A. 2006 Jul 7;1120(1-2):1-12. doi: 10.1016/j.chroma.2006.03.013. Epub 2006 Apr 4. PMID 16600255
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Juniper EF, Svensson K, Mork AC, Stahl E. Measurement properties and interpretation of three shortened versions of the asthma control questionnaire. Respir Med. 2005 May;99(5):553-8. doi: 10.1016/j.rmed.2004.10.008. Epub 2004 Nov 26. PMID 15823451
- [Background] Jurado C, Kintz P, Menendez M, Repetto M. Influence of the cosmetic treatment of hair on drug testing. Int J Legal Med. 1997;110(3):159-63. doi: 10.1007/s004140050056. PMID 9228567
- [Background] Kintz P. Value of the concept of minimal detectable dosage in human hair. Forensic Sci Int. 2012 May 10;218(1-3):28-30. doi: 10.1016/j.forsciint.2011.10.018. Epub 2011 Oct 20. PMID 22018745
- [Background] Kintz P, Alvarez JC, Deveaux M, Dumestre V, Gaillard Y, Gaulier JM. Conflicting hair testing results can have an impact in courts: interpretation of single exposure to zolpidem. J Anal Toxicol. 2014 Jun;38(5):304-5. doi: 10.1093/jat/bku014. Epub 2014 Mar 11. No abstract available. PMID 24618638
- [Background] Kintz P, Cirimele V, Ludes B. Pharmacological criteria that can affect the detection of doping agents in hair. Forensic Sci Int. 2000 Jan 10;107(1-3):325-34. doi: 10.1016/s0379-0738(99)00176-0. PMID 10689584
- [Background] Kintz P, Dumestre-Toulet V, Jamey C, Cirimele V, Ludes B. Doping control for beta-adrenergic compounds through hair analysis. J Forensic Sci. 2000 Jan;45(1):170-4. PMID 10641933
- [Background] Kronkvist K, Gustavsson M, Wendel AK, Jaegfeldt H. Automated sample preparation for the determination of budesonide in plasma samples by liquid chromatography and tandem mass spectrometry. J Chromatogr A. 1998 Oct 9;823(1-2):401-9. doi: 10.1016/s0021-9673(98)00592-5. PMID 9818417
- [Background] Kronstrand R, Ahlner J, Dizdar N, Larson G. Quantitative analysis of desmethylselegiline, methamphetamine, and amphetamine in hair and plasma from Parkinson patients on long-term selegiline medication. J Anal Toxicol. 2003 Apr;27(3):135-41. doi: 10.1093/jat/27.3.135. PMID 12731653
- [Background] Kronstrand R, Roman M, Hedman M, Ahlner J, Dizdar N. Dose-hair concentration relationship and pigmentation effects in patients on low-dose clozapine. Forensic Sci Med Pathol. 2007 Jun;3(2):107-14. doi: 10.1007/s12024-007-0010-9. Epub 2007 May 9. PMID 25869041
- [Background] LeBeau MA, Montgomery MA, Brewer JD. The role of variations in growth rate and sample collection on interpreting results of segmental analyses of hair. Forensic Sci Int. 2011 Jul 15;210(1-3):110-6. doi: 10.1016/j.forsciint.2011.02.015. Epub 2011 Mar 6. PMID 21382678
- [Background] Lee KM, Kim HJ, Son J, Park JH, Kwon OS, Lee J. Simple quantitation of formoterol and 11-nor-Delta(9)-tetrahydrocannabinol-9-carboxylic acid in human urine by liquid chromatography-tandem mass spectrometry in doping control. J Chromatogr B Analyt Technol Biomed Life Sci. 2014 Sep 15;967:8-12. doi: 10.1016/j.jchromb.2014.07.009. Epub 2014 Jul 14. PMID 25063922
- [Background] Lemaire-Hurtel, A.-S., Durand-Maugard, C., Berquin, P., Antonios, M., Hary, L., Andrejak, M., Masson, H., Manaouil, C., Abe, E. and Alvarez, J.-C. (2010).
- [Background] Li N, Tattam B, Brow KF, Seale JP. Quantification of epimeric budesonide and fluticasone propionate in human plasma by liquid chromatography-atmospheric pressure chemical ionization tandem mass spectrometry. J Chromatogr B Biomed Sci Appl. 2001 Sep 25;761(2):177-85. doi: 10.1016/s0378-4347(01)00329-2. PMID 11587347
- [Background] Li YN, Tattam B, Brown KF, Seale JP. Determination of epimers 22R and 22S of budesonide in human plasma by high-performance liquid chromatography-atmospheric pressure chemical ionization mass spectrometry. J Chromatogr B Biomed Appl. 1996 Aug 30;683(2):259-68. doi: 10.1016/0378-4347(96)00111-9. PMID 8891924
- [Background] Lindberg C, Blomqvist A, Paulson J. Determination of (22R,S)budesonide in human plasma by automated liquid chromatography/thermospray mass spectrometry. Biol Mass Spectrom. 1992 Nov;21(11):525-33. doi: 10.1002/bms.1200211102. PMID 1457467
- [Background] Liu AY, Yang Q, Huang Y, Bacchetti P, Anderson PL, Jin C, Goggin K, Stojanovski K, Grant R, Buchbinder SP, Greenblatt RM, Gandhi M. Strong relationship between oral dose and tenofovir hair levels in a randomized trial: hair as a potential adherence measure for pre-exposure prophylaxis (PrEP). PLoS One. 2014 Jan 8;9(1):e83736. doi: 10.1371/journal.pone.0083736. eCollection 2014. PMID 24421901
- [Background] Loussouarn G, Lozano I, Panhard S, Collaudin C, El Rawadi C, Genain G. Diversity in human hair growth, diameter, colour and shape. An in vivo study on young adults from 24 different ethnic groups observed in the five continents. Eur J Dermatol. 2016 Apr 1;26(2):144-54. doi: 10.1684/ejd.2015.2726. PMID 27019510
- [Background] Lu Y, Sun Z, Zhang Y, Chen X, Zhong D. Simultaneous quantification of 22R and 22S epimers of budesonide in human plasma by ultra-high-performance liquid chromatography-tandem mass spectrometry: application in a stereoselective pharmacokinetic study. J Chromatogr B Analyt Technol Biomed Life Sci. 2013 Mar 15;921-922:27-34. doi: 10.1016/j.jchromb.2013.01.015. Epub 2013 Jan 28. PMID 23416292
- [Background] Mancebo, M., Grassin-Delyle, S., Essid, A., Bataille, J., Guérard, P., Delyle, A. G. and Alvarez, J.-C. (2011).
- [Background] Mascher DG, Zech K, Nave R, Kubesch KM, Mascher HJ. Ultra-sensitive determination of Formoterol in human serum by high performance liquid chromatography and electrospray tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2006 Jan 2;830(1):25-34. doi: 10.1016/j.jchromb.2005.10.022. Epub 2005 Nov 7. PMID 16275132
- [Background] Mazzarino M, de la Torre X, Fiacco I, Pompei C, Calabrese F, Botre F. A simplified procedure for the analysis of formoterol in human urine by liquid chromatography-electrospray tandem mass spectrometry: application to the characterization of the metabolic profile and stability of formoterol in urine. J Chromatogr B Analyt Technol Biomed Life Sci. 2013 Jul 15;931:75-83. doi: 10.1016/j.jchromb.2013.05.021. Epub 2013 May 28. PMID 23777613
- [Background] Millar SE. Molecular mechanisms regulating hair follicle development. J Invest Dermatol. 2002 Feb;118(2):216-25. doi: 10.1046/j.0022-202x.2001.01670.x. PMID 11841536
- [Background] Miller-Larsson A, Mattsson H, Hjertberg E, Dahlback M, Tunek A, Brattsand R. Reversible fatty acid conjugation of budesonide. Novel mechanism for prolonged retention of topically applied steroid in airway tissue. Drug Metab Dispos. 1998 Jul;26(7):623-30. PMID 9660844
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Miramont S, Alvarez JC, Bourgogne E, Cheron G. [Passive cocaine inhalation by a 25-month-old child]. Arch Pediatr. 2013 Jun;20(6):654-6. doi: 10.1016/j.arcped.2013.03.006. Epub 2013 Apr 19. French. PMID 23608459
- [Background] Mortimer KJ, Harrison TW, Tang Y, Wu K, Lewis S, Sahasranaman S, Hochhaus G, Tattersfield AE. Plasma concentrations of inhaled corticosteroids in relation to airflow obstruction in asthma. Br J Clin Pharmacol. 2006 Oct;62(4):412-9. doi: 10.1111/j.1365-2125.2006.02712.x. PMID 16995862
- [Background] Nilsson K, Andersson M, Beck O. Phospholipid removal combined with a semi-automated 96-well SPE application for determination of budesonide in human plasma with LC-MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2014 Nov 1;970:31-5. doi: 10.1016/j.jchromb.2014.08.035. Epub 2014 Sep 6. PMID 25228411
- [Background] Noppe G, de Rijke YB, Dorst K, van den Akker EL, van Rossum EF. LC-MS/MS-based method for long-term steroid profiling in human scalp hair. Clin Endocrinol (Oxf). 2015 Aug;83(2):162-6. doi: 10.1111/cen.12781. Epub 2015 Apr 27. PMID 25823708
- [Background] Pecoraro, V. and Astore, I. P. L. (1990). Measurements of hair growth under physiological conditions. Hair and Hair Diseases. C. E. Orfanos and R. Happle. Berlin, Heidelberg, Springer Berlin Heidelberg: 237-254.
- [Background] Potsch L. A discourse on human hair fibers and reflections on the conservation of drug molecules. Int J Legal Med. 1996;108(6):285-93. doi: 10.1007/BF02432122. PMID 8793635
- [Background] Pragst F, Balikova MA. State of the art in hair analysis for detection of drug and alcohol abuse. Clin Chim Acta. 2006 Aug;370(1-2):17-49. doi: 10.1016/j.cca.2006.02.019. Epub 2006 Mar 6. PMID 16624267
- [Background] Pritchett JS, Phinney KW. Influence of chemical straightening on the stability of drugs of abuse in hair. J Anal Toxicol. 2015 Jan-Feb;39(1):13-6. doi: 10.1093/jat/bku106. Epub 2014 Oct 8. PMID 25298521
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Eur Respir J. 1993 Mar;6 Suppl 16:5-40. doi: 10.1183/09041950.005s1693. No abstract available. PMID 24576915
- [Background] Ray A, Raundhal M, Oriss TB, Ray P, Wenzel SE. Current concepts of severe asthma. J Clin Invest. 2016 Jul 1;126(7):2394-403. doi: 10.1172/JCI84144. Epub 2016 Jul 1. PMID 27367183
- [Background] Ribot M, Polito A, Grassin-Delyle S, Annane D, Alvarez JC. Human plasma quantification of fludrocortisone using liquid chromatography coupled with atmospheric pressure chemical ionization mass spectrometry after low-dosage administration. Clin Chim Acta. 2013 May;420:109-13. doi: 10.1016/j.cca.2012.11.026. Epub 2012 Dec 7. PMID 23228845
- [Background] Ricard F, Abe E, Duverneuil-Mayer C, Charlier P, de la Grandmaison G, Alvarez JC. Measurement of atropine and scopolamine in hair by LC-MS/MS after Datura stramonium chronic exposure. Forensic Sci Int. 2012 Nov 30;223(1-3):256-60. doi: 10.1016/j.forsciint.2012.09.015. Epub 2012 Oct 22. PMID 23084788
- [Background] Roberts JK, Cook SF, Stockmann C, Rollins DE, Wilkins DG, Sherwin CM. A Population Pharmacokinetic Analysis of Dextroamphetamine in the Plasma and Hair of Healthy Adults. Clin Drug Investig. 2015 Oct;35(10):633-43. doi: 10.1007/s40261-015-0323-5. PMID 26329917
- [Background] Rohrich J, Zorntlein S, Potsch L, Skopp G, Becker J. Effect of the shampoo Ultra Clean on drug concentrations in human hair. Int J Legal Med. 2000;113(2):102-6. doi: 10.1007/pl00007707. PMID 10741485
- [Background] Rollins DE, Wilkins DG, Krueger GG, Augsburger MP, Mizuno A, O'Neal C, Borges CR, Slawson MH. The effect of hair color on the incorporation of codeine into human hair. J Anal Toxicol. 2003 Nov-Dec;27(8):545-51. doi: 10.1093/jat/27.8.545. PMID 14670132
- [Background] Baque CS, Zhou J, Gu W, Collaudin C, Kravtchenko S, Kempf JY, Saint-Leger D. Relationships between hair growth rate and morphological parameters of human straight hair: a same law above ethnical origins? Int J Cosmet Sci. 2012 Apr;34(2):111-6. doi: 10.1111/j.1468-2494.2011.00687.x. Epub 2011 Oct 21. PMID 21951315
- [Background] Salomone A, Tsanaclis L, Agius R, Kintz P, Baumgartner MR. European guidelines for workplace drug and alcohol testing in hair. Drug Test Anal. 2016 Oct;8(10):996-1004. doi: 10.1002/dta.1999. Epub 2016 Jul 12. PMID 27402378
- [Background] Sardela VF, Deventer K, Pereira HM, de Aquino Neto FR, Van Eenoo P. Development and validation of a ultra high performance liquid chromatography-tandem mass spectrometric method for the direct detection of formoterol in human urine. J Pharm Biomed Anal. 2012 Nov;70:471-5. doi: 10.1016/j.jpba.2012.06.042. Epub 2012 Jul 7. PMID 22841556
- [Background] Skopp G, Potsch L, Moeller MR. On cosmetically treated hair--aspects and pitfalls of interpretation. Forensic Sci Int. 1997 Jan 17;84(1-3):43-52. doi: 10.1016/s0379-0738(96)02047-6. PMID 9042709
- [Background] Streel B, Cahay B, Klinkenberg R. Using total error concept for the validation of a liquid chromatography-tandem mass spectrometry method for the determination of budesonide epimers in human plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Aug 1;877(23):2290-300. doi: 10.1016/j.jchromb.2009.02.004. Epub 2009 Feb 11. PMID 19249257
- [Background] Sullivan SD, Rasouliyan L, Russo PA, Kamath T, Chipps BE; TENOR Study Group. Extent, patterns, and burden of uncontrolled disease in severe or difficult-to-treat asthma. Allergy. 2007 Feb;62(2):126-33. doi: 10.1111/j.1398-9995.2006.01254.x. PMID 17298420
- [Background] Szeitz A, Manji J, Riggs KW, Thamboo A, Javer AR. Validated assay for the simultaneous determination of cortisol and budesonide in human plasma using ultra high performance liquid chromatography-tandem mass spectrometry. J Pharm Biomed Anal. 2014 Mar;90:198-206. doi: 10.1016/j.jpba.2013.12.006. Epub 2013 Dec 16. PMID 24389462
- [Background] Taylor RL, Grebe SK, Singh RJ. Quantitative, highly sensitive liquid chromatography-tandem mass spectrometry method for detection of synthetic corticosteroids. Clin Chem. 2004 Dec;50(12):2345-52. doi: 10.1373/clinchem.2004.033605. Epub 2004 Oct 14. PMID 15486026
- [Background] Thevis M, Opfermann G, Schanzer W. Liquid chromatography/electrospray ionization tandem mass spectrometric screening and confirmation methods for beta2-agonists in human or equine urine. J Mass Spectrom. 2003 Nov;38(11):1197-206. doi: 10.1002/jms.542. PMID 14648827
- [Background] Thomas A, Geyer H, Schanzer W, Crone C, Kellmann M, Moehring T, Thevis M. Sensitive determination of prohibited drugs in dried blood spots (DBS) for doping controls by means of a benchtop quadrupole/Orbitrap mass spectrometer. Anal Bioanal Chem. 2012 May;403(5):1279-89. doi: 10.1007/s00216-011-5655-2. Epub 2012 Jan 10. PMID 22231507
- [Background] Thorsson L, Edsbacker S, Conradson TB. Lung deposition of budesonide from Turbuhaler is twice that from a pressurized metered-dose inhaler P-MDI. Eur Respir J. 1994 Oct;7(10):1839-44. doi: 10.1183/09031936.94.07101839. PMID 7828694
- [Background] Tosi A, Misciali C, Piraccini BM, Peluso AM, Bardazzi F. Drug-induced hair loss and hair growth. Incidence, management and avoidance. Drug Saf. 1994 Apr;10(4):310-7. doi: 10.2165/00002018-199410040-00005. PMID 8018303
- [Background] Tsanaclis L, Nutt J, Bagley K, Bevan S, Wicks J. Differentiation between consumption and external contamination when testing for cocaine and cannabis in hair samples. Drug Test Anal. 2014 Jun;6 Suppl 1:37-41. doi: 10.1002/dta.1623. PMID 24817047
- [Background] van den Brink KI, Boorsma M, Staal-van den Brekel AJ, Edsbacker S, Wouters EF, Thorsson L. Evidence of the in vivo esterification of budesonide in human airways. Br J Clin Pharmacol. 2008 Jul;66(1):27-35. doi: 10.1111/j.1365-2125.2008.03164.x. Epub 2008 Apr 1. PMID 18384442
- [Background] Van Neste D. Thickness, medullation and growth rate of female scalp hair are subject to significant variation according to pigmentation and scalp location during ageing. Eur J Dermatol. 2004 Jan-Feb;14(1):28-32. PMID 14965792
- [Background] Van Neste D. Why care about linear hair growth rates (LHGR)? a study using in vivo imaging and computer assisted image analysis after manual processing (CAIAMP) in unaffected male controls and men with male pattern hair loss (MPHL). Eur J Dermatol. 2014 Sep-Oct;24(5):568-76. doi: 10.1684/ejd.2014.2428. PMID 25445091
- [Background] Van Neste DJ, Rushton DH. Gender differences in scalp hair growth rates are maintained but reduced in pattern hair loss compared to controls. Skin Res Technol. 2016 Aug;22(3):363-9. doi: 10.1111/srt.12274. Epub 2015 Nov 3. PMID 26526232
- [Background] van Zyl GU, van Mens TE, McIlleron H, Zeier M, Nachega JB, Decloedt E, Malavazzi C, Smith P, Huang Y, van der Merwe L, Gandhi M, Maartens G. Low lopinavir plasma or hair concentrations explain second-line protease inhibitor failures in a resource-limited setting. J Acquir Immune Defic Syndr. 2011 Apr;56(4):333-9. doi: 10.1097/QAI.0b013e31820dc0cc. PMID 21239995
- [Background] Wang Y, Tang Y, Moellmann H, Hochhaus G. Simultaneous quantification of budesonide and its two metabolites, 6beta-hydroxybudesonide and 16alpha-hydroxyprednisolone, in human plasma by liquid chromatography negative electrospray ionization tandem mass spectrometry. Biomed Chromatogr. 2003 Mar-Apr;17(2-3):158-64. doi: 10.1002/bmc.233. PMID 12717805
- [Background] Wenzel SE. Complex phenotypes in asthma: current definitions. Pulm Pharmacol Ther. 2013 Dec;26(6):710-5. doi: 10.1016/j.pupt.2013.07.003. Epub 2013 Jul 20. PMID 23880027
- [Background] Williams J, Patsalos PN, Mei Z, Schapel G, Wilson JF, Richens A. Relation between dosage of carbamazepine and concentration in hair and plasma samples from a compliant inpatient epileptic population. Ther Drug Monit. 2001 Feb;23(1):15-20. doi: 10.1097/00007691-200102000-00004. PMID 11206037
- [Background] Yegles M, Marson Y, Wennig R. Influence of bleaching on stability of benzodiazepines in hair. Forensic Sci Int. 2000 Jan 10;107(1-3):87-92. doi: 10.1016/s0379-0738(99)00152-8. PMID 10689563